CLINICAL TRIAL: NCT01874054
Title: A Phase 1/2 Single-arm, Open-label Study to Evaluate the Safety and Efficacy of Brentuximab Vedotin in Combination With Bendamustine in Patients With Relapsed or Refractory Hodgkin Lymphoma (HL)
Brief Title: Study of Brentuximab Vedotin Combined With Bendamustine in Patients With Hodgkin Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGN35-016
Record Dates: First submitted 2013-06-06; First posted 2013-06-10 (Estimated); Results first posted 2017-04-06 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-01

CONDITIONS: Hodgkin Disease
Keywords: Antibody-Drug Conjugate; Antibodies, Monoclonal; Hodgkin Disease; Hematologic Diseases; Drug Therapy; Immunotherapy; Antigens, CD30; Lymphoma; monomethylauristatin E
MeSH Terms: conditions — Hodgkin Disease; Hematologic Diseases; Lymphoma | interventions — Brentuximab Vedotin; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Brentuximab Vedotin + Bendamustine (Experimental): Brentuximab vedotin 1.8 mg/kg every 3 weeks for up to 16 cycles by IV infusion and bendamustine 90 mg/m2 on Days 1 and 2 every 3 weeks by IV infusion for up to 6 cycles
  Interventions: Drug: brentuximab vedotin; Drug: bendamustine

INTERVENTIONS:
Drug: brentuximab vedotin — 1.8 mg/kg every 3 weeks by intravenous (IV) infusion
  Other Names: Adcetris; SGN-35
Drug: bendamustine — 90 mg/m2 on Days 1 and 2 of 3-week cycles

SUMMARY:
The purpose of this study is to assess safety and efficacy of brentuximab vedotin in combination with bendamustine in patients with relapsed or refractory Hodgkin lymphoma. It is an open-label, 2-stage study designed to determine the recommended dose level of bendamustine in combination with brentuximab vedotin. The study will assess the safety profile of the combination treatment and determine what proportion of patients achieve a complete remission.

ELIGIBILITY:
Inclusion Criteria:

* Histopathological diagnosis of classical Hodgkin lymphoma
* Failed standard front-line therapy
* Measurable disease of at least 1.5 cm as documented by radiographic technique
* Eastern Cooperative Oncology Group performance status less than or equal to 2

Exclusion Criteria:

* Received prior salvage therapy, including radiotherapy
* Chemotherapy, radiotherapy, biologics, and/or other treatment with immunotherapy not completed 4 weeks prior to first dose of study drug
* Concurrent use of other investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2013-06; Primary Completion 2015-12 (Actual); Study Completion 2018-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil Josephson, MD, Study Director — Seagen Inc.
Locations (13):
- United States (13):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Pacific Hematology Oncology Associates, San Francisco, California
  - Stanford Cancer Center, Stanford, California
  - Oncology Institute of Hope & Innovation, The, Whittier, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic Minnesota, Rochester, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Columbia University Medical Center, New York, New York
  - Jewish Hospital, The, Cincinnati, Ohio
  - Case Western Reserve University / University Hospitals Case Medical Center, Cleveland, Ohio
  - Saint Francis Hospital / Bon Secours, Greenville, South Carolina
  - Charles A. Sammons Cancer Center / Baylor University Medical Center, Dallas, Texas

REFERENCES:
- [Derived] LaCasce AS, Bociek RG, Sawas A, Caimi P, Agura E, Matous J, Ansell SM, Crosswell HE, Islas-Ohlmayer M, Behler C, Cheung E, Forero-Torres A, Vose J, O'Connor OA, Josephson N, Wang Y, Advani R. Brentuximab vedotin plus bendamustine: a highly active first salvage regimen for relapsed or refractory Hodgkin lymphoma. Blood. 2018 Jul 5;132(1):40-48. doi: 10.1182/blood-2017-11-815183. Epub 2018 Apr 27. PMID 29703778

RESULTS

PARTICIPANT FLOW:
Recruitment Details: June 2013 - July 2016
Groups:
- Brentuximab Vedotin + Bendamustine: brentuximab vedotin (BV): 1.8 mg/kg on Day 1 of 3-week cycles by intravenous (IV) infusion
  bendamustine: 90 mg/m^2 on Days 1 and 2 of 3-week cycles by intravenous (IV) infusion
Period: Overall Study
Arm/Group | Brentuximab Vedotin + Bendamustine
Started | 55
Completed ≥2 Cycles of Combo Treatment | 53
Completed 16 Cycles of BV Treatment | 17
Completed (No patients completed per protocol as there was no pre-defined follow-up period) | 0
Not Completed | 55
Not completed — Withdrawal by Subject | 3
Not completed — Study Termination by Sponsor | 42
Not completed — Lost to Follow-up | 5
Not completed — Death | 5

BASELINE CHARACTERISTICS:
Population: All subjects who enrolled and received at least 1 dose of brentuximab vedotin.
Groups:
- Brentuximab Vedotin + Bendamustine: brentuximab vedotin: 1.8 mg/kg on Day 1 of 3-week cycles by intravenous (IV) infusion
  bendamustine: 90 mg/m^2 on Days 1 and 2 of 3-week cycles by intravenous (IV) infusion
Arm/Group | Brentuximab Vedotin + Bendamustine
Number analyzed (Participants) | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 50
  >=65 years | 5
Age, Continuous [Median (Full Range); unit: years] | 36 [19 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 51
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 46
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 55
Eastern Cooperative Group Oncology Performance Status [Count of Participants; unit: Participants] — 0=Normal activity; 1=Symptoms but ambulatory; 2=In bed <50% of the time; 3= In bed >50% of the time; 4=100% bedridden; 5=Dead
  Participants
    0 | 31
    1 | 23
    2 | 1

OUTCOME MEASURES:

1. Primary Outcome: Complete Remission Rate
Description: Complete remission rate among all subjects (Phase 1 and 2 combined) treated at the dose level selected for Phase 2. Complete remission (CR) per Cheson 2007 Revised Response Criteria for Malignant Lymphoma is a disappearance of all evidence of disease.
Time Frame: Up to 4.6 months
Population: All patients who received at least 2 cycles of combination treatment at the recommended dose level and had a baseline tumor assessment and at least 1 postbaseline tumor assessment, or who had documented disease progression (including clinical disease progression) at any time after the first dose of combination therapy at the recommended dose level.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Brentuximab Vedotin + Bendamustine
Number analyzed (Participants) | 53
percentage of participants | 73.6 [59.67 to 84.74]

2. Primary Outcome: Incidence of Adverse Events (AEs)
Description: All AEs reported after initiation of treatment and pre-existing conditions that worsen after initiation of treatment will be considered treatment-emergent AEs (TEAEs). All AEs will be coded by system organ class, MedDRA preferred term, and severity grade using NCI CTCAE V4.03. All recorded AEs will be included in the data listings.
Time Frame: Up to 13.8 months
Population: All subjects who were enrolled and received at least 1 dose of brentuximab vedotin.
Measure: Count of Participants; unit: Participants
Arm/Group | Brentuximab Vedotin + Bendamustine
Number analyzed (Participants) | 55
Participants
  Any Treatment-Emergent Adverse Event (TEAE) | 55
  Any TEAE with Severity >= Grade 3 | 31
  Any Treatment-Related Adverse Event | 54
  Any Serious Adverse Event | 18
  Any Treatment-Related Serious Adverse Event | 15
  Treatment Discontinuation Due to Adverse Event | 20

3. Secondary Outcome: Incidence of Dose-limiting Toxicities
Description: Incidence of dose-limiting toxicity (DLT) was evaluated in an initial safety cohort of 10 patients who were followed for protocol-defined DLT events until Cycle 2 Day 1.
Time Frame: Up to 3 weeks; first cycle of therapy through the first day of Cycle 2
Population: An initial safety cohort of 10 patients who enrolled and received at least 1 dose of brentuximab vedotin were evaluated for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Brentuximab Vedotin + Bendamustine
Number analyzed (Participants) | 10
Participants | 0

4. Secondary Outcome: Overall Best Response Rate
Description: Percentage of participants who achieved a best response of complete remission (CR, disappearance of all evidence of disease), partial remission (PR, regression of greater than or equal to 50% of measurable disease and no new sites), stable disease (SD, failure to obtain a complete or partial response or progressive disease), or progressive disease (PD, any new lesion or increase by 50% or more of previously involved sites from nadir) per Cheson 2007 Revised Response Criteria for Malignant Lymphoma
Time Frame: Up to 4.6 months
Population: All patients who received at least 2 cycles of combination treatment, had a baseline tumor assessment, and at least 1 post-baseline tumor assessment, or who had documented disease progression (including clinical disease progression) any time after the first dose of combination therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Brentuximab Vedotin + Bendamustine
Number analyzed (Participants) | 53
Participants
  Complete Remission | 39
  Partial Remission | 10
  Stable Disease | 3
  Progressive Disease | 1

5. Secondary Outcome: Duration of Response
Description: The time from first observation of remission to disease progression/relapse or death from any cause, whichever occurs first.
Time Frame: Up to 47.8 months
Population: Patients with a complete or partial response who received at least 2 cycles of combination treatment and had a baseline tumor assessment and at least 2 post-baseline tumor assessment, or who had documented disease progression (including clinical disease progression) at any time after the first dose of combination therapy.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Brentuximab Vedotin + Bendamustine
Number analyzed (Participants) | 49
months | 43.0 [18.7 to 47.8]

6. Secondary Outcome: Progression-free Survival
Description: The time from first dose of study medication to first documentation of disease progression/relapse, or to death due to any cause, whichever occurs first.
Time Frame: Up to 49 months
Population: All patients who received at least 2 cycles of combination treatment and had a baseline tumor assessment and at least 1 post-baseline tumor assessment, or who had documented disease progression (including clinical disease progression) at any time after the first dose of combination therapy.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Brentuximab Vedotin + Bendamustine
Number analyzed (Participants) | 53
months | 44.2 [20.9 to 49.0]

ADVERSE EVENTS:
Time Frame: Up to 13.8 months
Description: Treatment-emergent adverse events: a newly occurring or worsening adverse event after the first dose of study drug.
Arm/Group | Brentuximab Vedotin + Bendamustine
All-Cause Mortality (participants affected / at risk) | 5/55
Serious Adverse Events (participants affected / at risk) | 18/55
Other Adverse Events (participants affected / at risk) | 55/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brentuximab Vedotin + Bendamustine (N=55)
Pyrexia (General disorders) | 8
Chills (General disorders) | 3
Malaise (General disorders) | 2
Pain (General disorders) | 1
Hypotension (Vascular disorders) | 5
Deep vein thrombosis (Vascular disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Colitis (Gastrointestinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Urticaria (Skin and subcutaneous tissue disorders) | 2
Erythema (Skin and subcutaneous tissue disorders) | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Phlebitis infective (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Syncope (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brentuximab Vedotin + Bendamustine (N=55)
Nausea (Gastrointestinal disorders) | 40
Diarrhoea (Gastrointestinal disorders) | 20
Vomiting (Gastrointestinal disorders) | 20
Constipation (Gastrointestinal disorders) | 17
Abdominal pain (Gastrointestinal disorders) | 5
Dry mouth (Gastrointestinal disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 4
Dysphagia (Gastrointestinal disorders) | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3
Fatigue (General disorders) | 30
Chills (General disorders) | 15
Pyrexia (General disorders) | 15
Oedemia peripheral (General disorders) | 7
Pain (General disorders) | 7
Malaise (General disorders) | 4
Non-cardiac chest pain (General disorders) | 4
Asthenia (General disorders) | 3
Chest discomfort (General disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 14
Rash (Skin and subcutaneous tissue disorders) | 14
Pruritus (Skin and subcutaneous tissue disorders) | 13
Rash generalised (Skin and subcutaneous tissue disorders) | 7
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7
Rash pruritic (Skin and subcutaneous tissue disorders) | 6
Night sweats (Skin and subcutaneous tissue disorders) | 5
Erythema (Skin and subcutaneous tissue disorders) | 3
Pruritus generalised (Skin and subcutaneous tissue disorders) | 3
Rash erythematous (Skin and subcutaneous tissue disorders) | 3
Swelling face (Skin and subcutaneous tissue disorders) | 3
Peripheral sensory neuropathy (Nervous system disorders) | 14
Headache (Nervous system disorders) | 11
Neuropathy peripheral (Nervous system disorders) | 10
Dizziness (Nervous system disorders) | 8
Paraesthesia (Nervous system disorders) | 8
Hypoaesthesia (Nervous system disorders) | 4
Dysgeusia (Nervous system disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 13
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 5
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 3
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 10
Bone pain (Musculoskeletal and connective tissue disorders) | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 8
Muscular weakness (Musculoskeletal and connective tissue disorders) | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 3
Decreased appetite (Metabolism and nutrition disorders) | 10
Dehydration (Metabolism and nutrition disorders) | 5
Hypokalaemia (Metabolism and nutrition disorders) | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 4
Hyperuricaemia (Metabolism and nutrition disorders) | 3
Flushing (Vascular disorders) | 10
Hot flush (Vascular disorders) | 6
Hypotension (Vascular disorders) | 3
Upper respiratory tract infection (Infections and infestations) | 8
Urinary tract infection (Infections and infestations) | 5
Herpes zoster (Infections and infestations) | 3
Weight decreased (Investigations) | 5
Lymphopenia (Blood and lymphatic system disorders) | 7
Neutropenia (Blood and lymphatic system disorders) | 4
Insomnia (Psychiatric disorders) | 11
Anxiety (Psychiatric disorders) | 5
Tachycardia (Cardiac disorders) | 3
Ear pain (Ear and labyrinth disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 18 months after conclusion or termination of a study at all sites. After such multi-site publication, all proposed site publications and presentations will be submitted to the Sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.